CLINICAL TRIAL: NCT01444209
Title: Interstitial Radioactive Iodine Implants for the Treatment of Pan-invasive Pituitary Macroadenomas
Brief Title: Radioactive Iodine Implants for Pan-invasive Pituitary Macroadenomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to accrue
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 042011-075
Record Dates: First submitted 2011-09-22; First posted 2011-09-30 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Pituitary Macroadenoma
Keywords: pituitary gland
MeSH Terms: conditions — Pituitary Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Therapy (Experimental): Interstitial Radioactive Iodine Implants
  Interventions: Radiation: Iodine Implants

INTERVENTIONS:
Radiation: Iodine Implants — Interstitial Radioactive Iodine Implants

SUMMARY:
This study is a single arm Phase II pilot trial. Patients enrolled on the trial will undergo implantation of high activity iodine-125 seeds into their pituitary adenoma. The tumor response to treatment will be monitored as well as change in visual fields, associated adverse effects, progression free survival and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pathological or radiographic diagnosis of a pan-invasive pituitary macroadenoma
* Pan-invasive for the purposes of the protocol will be defined as meeting each of the following 2 major criteria: (1). tumor volume greater than 20 cc at enrollment, and (2). suprasellar extension. In addition, a pan-invasive tumor must meet any one of the following 3 minor criteria, a) unresectable tumor invasion into a cavernous sinus, b) bone or bone marrow invasion into the clivus or temporal bones, or c) tumor extension in any direction unlikely to be completely removed by specifically a transphenoidal surgical approach.
* Patients who meet the two major criteria above (1 and 2) and are medically inoperable for tumor resection (due to confounding co-existing medical problems) are eligible without meeting any of the three minor criteria (a, b, or c).
* Patients should be immediately threatened for vision loss or other significant neurological impairment directly related to tumor mass effect. As such, all patients enrolled would likely benefit from tumor response (shrinkage).
* Patients must have visible tumor on imaging studies (MRI or CT)
* The patient's Zubrod performance status must be 0-3.
* Patients must be at least 18 years of age.
* Mandatory Imaging Studies: Must be done 45 or fewer days prior to :

MRI or CT scan of the brain including the entire skull base and all areas of tumor extension

Exclusion Criteria:

* Patients who are unable to undergo general anesthesia
* Patients who are unable to undergo placement of a stereotactic head frame
* Patients who are unable to provide informed consent
* Patients who are pregnant or nursing
* Patients with severe kidney dysfunction
* Patients who have contraindications to MRI, such as implanted pacemaker device
* Patients with diagnosis of pituitary carcinoma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Timmerman, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Partial Response (Reduction in 30% of Tumor Volume) or Greater Response Within 12 Months From the Implant Procedure.
Time Frame: 12 months
Population: No data collected
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Change of the Patient's Humphrey Visual Field Testing
Time Frame: 5 years
Population: Data were not collected
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Potential Toxicities Associated With Interstitial Seed Placement
Time Frame: 5 years
Population: No data collected
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival
Time Frame: 5 years
Population: No data collected
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: The Effect of the Treatment on Quality of Life Evaluations (Patient Reported Outcomes)
Time Frame: 5 years
Population: No data collected
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: The Cost-utility of the Treatment Arm (in Terms of the Primary Outcome) in Comparison With Other Widely Accepted Cancer and Non-cancer Therapies
Time Frame: 5 years
Population: No data collected
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: No data collected
Description: Data were not collected
Arm/Group | Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to failure to accrue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT01444209/Prot_SAP_000.pdf